CLINICAL TRIAL: NCT07115030
Title: Project STRONGER: Stepped Care for Opioid Use Disorder Treatment Engagement and Recovery
Acronym: STRONGER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000040103; R61DA059895 (NIH)
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-08

CONDITIONS: Opioid Use Disorder; Intimate Partner Violence (IPV); Post Traumatic Stress Disorder PTSD
Keywords: opioid use disorder; intimate partner violence; domestic violence
MeSH Terms: conditions — Opioid-Related Disorders; Combat Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCT+2HOPE (Experimental): During the first 12 weeks, participants will be offered PCT+ via eight 1-hour group sessions facilitated by a trained counselor ("facilitator") at the treatment program where they receive MOUD. The purpose of this group is to help participants address problems in their daily lives that arise from PTSD-related impairment in psychosocial functioning. After 12 weeks, participants who meet any of the following criteria will be "stepped up" to HOPE: 1) are not retained in MOUD treatment or 2) have moderate or higher impairment in PTSD-related psychosocial functioning. Participants who are "stepped up" will be offered 10 1-hour individual sessions over the next 14 weeks. HOPE is an individual counseling program designed for women in treatment for their opioid use, who have experienced abuse from an intimate partner and are experiencing PTSD-related impairment in psychosocial functioning.
  Interventions: Behavioral: PCT+2HOPE
- Treatment as Usual (No Intervention): Participants will be provided with a list of community resources and a referral to a local domestic violence service provider that can help address experiences of relationship strain with an intimate or romantic partner.

INTERVENTIONS:
Behavioral: PCT+2HOPE — Each PCT+ group follows the same structure and starts with the group setting an agenda. Clients identify issues to work on using these steps: 1) Identify an issue and if/how it relates to their PTSD or substance use, 2) Brainstorm ideas that may help, 3) Evaluate how useful each idea is, and 4) Choose a plan. Clients are encouraged to implement and evaluate the effectiveness of the plan and share the outcome at their next group. At the end of the group, clients process their experiences of the discussion.
  HOPE is a flexible, module-based individual treatment where the ordering and emphasis of each module are determined by client priorities. HOPE is trauma-focused; clients relate their current symptoms to their experience of IPV, but do not process traumatic memories. Modules focus on 1) Establishing safety, providing information and skills that enhance empowerment, 2) Cognitive behavioral therapy skills, and 3) Improving relationships and establishing healthy boundaries.
  Arms: PCT+2HOPE

SUMMARY:
Using a hybrid type 1 effectiveness-implementation approach, this study aims to evaluate the impact of a novel stepped care model ("PCT+2HOPE") versus treatment as usual (TAU) on increasing retention in community-based medication for opioid use disorder (MOUD) treatment among women who have experienced intimate partner violence (W-IPV). PCT+2HOPE includes Present-Centered Therapy (PCT+) with stepped care as indicated by moderate, severe, or extreme PTSD-related impairment in psychosocial functioning to Helping to Overcome PTSD through Empowerment (HOPE), two evidence-based behavioral interventions adapted for women with opioid use disorder (OUD). We will examine the effectiveness of PCT+2HOPE vs. TAU on the primary outcome (i.e., retention in MOUD treatment) and secondary outcomes related to trauma (i.e., PTSD-related impairment in psychosocial functioning and depression), substance use (i.e. OUD symptom severity, extra-medical opioid use [i.e., use of prescription opioids without a doctor's prescription; in greater amounts, more often, longer than prescribed, or for a reason other than a doctor said they should be used], and recovery), and empowerment. We will explore the extent to which the effectiveness of PCT+2HOPE vs. treatment as usual differs based on access to basic needs. We will also conduct an implementation-focused process evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Woman;
* Are ≥ 18 years old;
* Receive MOUD treatment at one of the participating sites;
* Have received MOUD for >14 days to allow for initial stabilization;
* Have initiated the current treatment episode within the past 12 months;
* Experienced physical or psychological IPV in their lifetime;
* Have at least moderate impairment in psychosocial functioning (on B-IPF) as a result of PTSD symptoms;
* Available during the date/time of the intervention group
* Able to read/understand English; and
* Provide written informed consent.

Exclusion Criteria:

* Fail a capacity-to-consent questionnaire;
* Have an unstable medical condition (e.g., hospitalization, planned surgery, newly starting chemotherapy, plans for palliative care) and/or unstable psychiatric illness (e.g., untreated psychosis) that would interfere with their ability to participate in study activities;
* Will be unavailable for >4 consecutive weeks during the study period (e.g., anticipated move, planned surgery);
* Are unable to read/understand English;
* Inability to provide at least one form of contact

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Retention in MOUD treatment | Week 26
  Retention in MOUD treatment at week 26. This will be measured through a combination of self-report with objective confirmation (e.g., via electronic health record, provider-confirmed treatment engagement/retention, medication bottles, urine toxicology testing).

SECONDARY OUTCOMES:
PTSD-related impairment in psychosocial functioning | Week 26
  The Brief-Inventory of Psychosocial Functioning (B-IPF) will be collected to assess PTSD-related impairment in functioning. The PCL-5 will be administered immediately prior and B-IPF items will be anchored to endorsed PTSD). B-IPF total scores represent an index of overall functional impairment, with higher scores indicating greater functional impairment.
Opioid use disorder symptom severity | Week 26
  Past 30-day opioid use disorder (OUD) symptom severity will be assessed with the Opioid Use Disorder Checklist, an 11-item assessment of DSM-5 criteria. DSM-5 considers 2 to 3 criteria mild; 4 to 5, moderate; and 6 to 11, severe OUD.
Days of extra-medical opioid use, past 30 days | Week 26
  Past 30-day opioid use will be assessed with the timeline follow back (TLFB) method to capture the number of days of extra-medical opioid use.
Urine test positive for opioid use | Week 26
  Urine toxicology testing will be performed to assess for the presence of extra-medical opioid use (e.g., opiates, oxycodone, fentanyl).
Depression symptom severity | Week 26
  The 9-item Patient Health Questionnaire (PHQ-9) will be collected to measure the prevalence and severity of the 9 DSM criteria for depression. The PHQ-9 uses a continuous score with higher scores indicating greater depression symptom severity and a 5-point change indicating clinically significant change.
Recovery | Week 26
  The 21-item Substance Use Recovery Evaluator (SURE) will be collected to measure substance use recovery. The SURE uses a continuous total recovery score between 21 and 63, with higher scores indicating "higher recovery scores."
Empowerment | Week 26
  The Personal Progress Scale-Revised (PPS-R) will be collected to measure empowerment. The PPS-R uses a continuous score with higher scores indicating higher empowerment.

CONTACTS AND LOCATIONS:
Overall Officials: Tami Sullivan, PhD, Principal Investigator — Yale University; E. Jennifer Edelman, MD, MHS, AAHIVS, Principal Investigator — Yale University; Dawn Johnson, PhD, Principal Investigator — The University of Akron
Locations (3):
- United States (3):
  - Liberation Programs, Bridgeport, Connecticut
  - Community Health Resources (CHR) Pathways Opiate Treatment Program, Enfield, Connecticut
  - The APT Foundation, Inc., West Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data and associated documentation will be made available to the research community free of charge through the Inter-university Consortium for Political and Social Research (ICPSR), which has been approved as a HEAL-compliant data repository.
Time Frame: Final submission and release of the study data will occur before the end of the award period. Study data deposited with ICPSR will be available to the research community in perpetuity. Datasets underlying methodological publications will be shared at or prior to initial publication date.

REFERENCES:
- [Background] Johnson DM, Zlotnick C, Gonzalez A. Treatment of Post-traumatic Stress Disorder in Survivors of Intimate Partner Violence. Handbook of Interpersonal Violence and Abuse Across the Lifespan: A project of the National Partnership to End Interpersonal Violence Across the Lifespan (NPEIV). 2021:3223-3246.
- [Background] Moullin JC, Dickson KS, Stadnick NA, Rabin B, Aarons GA. Systematic review of the Exploration, Preparation, Implementation, Sustainment (EPIS) framework. Implement Sci. 2019 Jan 5;14(1):1. doi: 10.1186/s13012-018-0842-6. PMID 30611302
- [Background] Morse AK, Sercombe J, Askovic M, Fisher A, Marel C, Chatterton ML, Kay-Lambkin F, Barrett E, Sunderland M, Harvey L, Peach N, Teesson M, Mills KL. Systematic review of the efficacy, effectiveness, and cost-effectiveness of stepped-care interventions for the prevention and treatment of problematic substance use. J Subst Abuse Treat. 2023 Jan;144:108928. doi: 10.1016/j.jsat.2022.108928. Epub 2022 Nov 4. PMID 36370469
- [Background] Carroll KM, Weiss RD. The Role of Behavioral Interventions in Buprenorphine Maintenance Treatment: A Review. Focus (Am Psychiatr Publ). 2019 Apr;17(2):183-192. doi: 10.1176/appi.focus.17206. Epub 2019 Apr 10. PMID 32021588
- [Background] Johnson DM, Johnson NL, Perez SK, Palmieri PA, Zlotnick C. Comparison of Adding Treatment of PTSD During and After Shelter Stay to Standard Care in Residents of Battered Women's Shelters: Results of a Randomized Clinical Trial. J Trauma Stress. 2016 Aug;29(4):365-73. doi: 10.1002/jts.22117. Epub 2016 Jul 26. PMID 27459503
- [Background] Johnson DM, Palmieri PA, Zlotnick C, Johnson NL, Hoffman L, Holmes SC, Ceroni TL. A Randomized Controlled Trial Comparing HOPE Treatment and Present-Centered Therapy in Women Residing in Shelter with PTSD from Intimate Partner Violence. Psychol Women Q. 2020 Dec 1;44(4):539-553. doi: 10.1177/0361684320953120. Epub 2020 Sep 17. PMID 34305273
- [Background] Schnurr PP, Friedman MJ, Engel CC, Foa EB, Shea MT, Chow BK, Resick PA, Thurston V, Orsillo SM, Haug R, Turner C, Bernardy N. Cognitive behavioral therapy for posttraumatic stress disorder in women: a randomized controlled trial. JAMA. 2007 Feb 28;297(8):820-30. doi: 10.1001/jama.297.8.820. PMID 17327524
- [Background] Belsher BE, Beech E, Evatt D, Smolenski DJ, Shea MT, Otto JL, Rosen CS, Schnurr PP. Present-centered therapy (PCT) for post-traumatic stress disorder (PTSD) in adults. Cochrane Database Syst Rev. 2019 Nov 18;2019(11):CD012898. doi: 10.1002/14651858.CD012898.pub2. PMID 31742672
- [Background] Butner JL, Gupta N, Fabian C, Henry S, Shi JM, Tetrault JM. Onsite treatment of HCV infection with direct acting antivirals within an opioid treatment program. J Subst Abuse Treat. 2017 Apr;75:49-53. doi: 10.1016/j.jsat.2016.12.014. Epub 2017 Jan 24. PMID 28237054
- [Background] Ngo BV, James JR, Blalock KL, Jackson SL, Chew LD, Tsui JI. Hepatitis C treatment outcomes among patients treated in co-located primary care and addiction treatment settings. J Subst Abuse Treat. 2021 Dec;131:108438. doi: 10.1016/j.jsat.2021.108438. Epub 2021 Apr 29. PMID 34098298
- [Background] Oldfield BJ, Munoz N, McGovern MP, Funaro M, Villanueva M, Tetrault JM, Edelman EJ. Integration of care for HIV and opioid use disorder. AIDS. 2019 Apr 1;33(5):873-884. doi: 10.1097/QAD.0000000000002125. PMID 30882491
- [Background] Bailey K, Trevillion K, Gilchrist G. What works for whom and why: A narrative systematic review of interventions for reducing post-traumatic stress disorder and problematic substance use among women with experiences of interpersonal violence. J Subst Abuse Treat. 2019 Apr;99:88-103. doi: 10.1016/j.jsat.2018.12.007. Epub 2018 Dec 24. PMID 30797400
- [Background] Sullivan TP, Armeli S, Tennen H, Weiss NH, Hansen NB. Fluctuations in daily PTSD symptoms are related to proximal alcohol use: a micro-longitudinal study of women victims of intimate partner violence. Am J Drug Alcohol Abuse. 2020;46(1):98-108. doi: 10.1080/00952990.2019.1624765. Epub 2019 Jul 16. PMID 31311330
- [Background] Sullivan TP, Cavanaugh CE, Buckner JD, Edmondson D. Testing posttraumatic stress as a mediator of physical, sexual, and psychological intimate partner violence and substance problems among women. J Trauma Stress. 2009 Dec;22(6):575-84. doi: 10.1002/jts.20474. PMID 19960546
- [Background] Hellmuth JC, Jaquier V, Swan SC, Sullivan TP. Elucidating posttraumatic stress symptom profiles and their correlates among women experiencing bidirectional intimate partner violence. J Clin Psychol. 2014 Oct;70(10):1008-21. doi: 10.1002/jclp.22100. Epub 2014 Apr 19. PMID 24752965
- [Background] Sullivan TP, Weiss NH, Price C, Pugh N, Hansen NB. Strategies for coping with individual PTSD symptoms: Experiences of African American victims of intimate partner violence. Psychol Trauma. 2018 May;10(3):336-344. doi: 10.1037/tra0000283. Epub 2017 May 8. PMID 28481562
- [Background] Peirce JM, Brooner RK, King VL, Kidorf MS. Effect of traumatic event reexposure and PTSD on substance use disorder treatment response. Drug Alcohol Depend. 2016 Jan 1;158:126-31. doi: 10.1016/j.drugalcdep.2015.11.006. Epub 2015 Nov 21. PMID 26652898
- [Background] Engstrom M, El-Bassel N, Gilbert L. Childhood sexual abuse characteristics, intimate partner violence exposure, and psychological distress among women in methadone treatment. J Subst Abuse Treat. 2012 Oct;43(3):366-76. doi: 10.1016/j.jsat.2012.01.005. Epub 2012 Mar 22. PMID 22444420